CLINICAL TRIAL: NCT05860608
Title: Multidisciplinary Approach for High-risk Patients Leading to Early Diagnosis of Canadians With Heart Failure.
Acronym: MAPLE-CHF
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: already submitted on NCT05859048
Sponsor: Montreal Heart Institute (Other)
Responsible Party: Principal Investigator, Anique Ducharme, MD, MSc. Professor of Medicine, Université de Montréal. Department of Medicine, Montreal Heart Institute, Montreal Heart Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023-001
Record Dates: First submitted 2023-05-08; First posted 2023-05-16 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ACTIVE investigational arm (NT-proBNP + AI-ECHO) (Experimental): NT-proBNP will be performed in all individuals randomized to the ACTIVE arm at the same visit as informed consent; those with elevated NT-proBNP (≥125pg/ml) will undergo an Us2.ai (AI-enabled report) handheld echocardiogram within one month of NT-proBNP testing. A standard echocardiographic study will be performed if the AI-echo is non-diagnostic.
  Interventions: Device: Us2.ai (AI-enabled report) handheld echocardiogram
- CONTROL routine care arm (Other): Patients randomized to usual care will undergo standard clinical follow-up, with NT-proBNP and conventional echocardiography prescribed only as per usual practice.
  Interventions: Device: Us2.ai (AI-enabled report) handheld echocardiogram

INTERVENTIONS:
Device: Us2.ai (AI-enabled report) handheld echocardiogram — NT-proBNP will be performed in all individuals randomized to the ACTIVE arm at the same visit as informed consent, and those with elevated NT-proBNP (≥125pg/ml) will be invited to attend a visit for an Us2.ai (AI-enabled) echocardiogram which will be controlled with a standard echocardiographic study if the AI-echo is non-diagnostic.

SUMMARY:
In the MAPLE-CHF trial, patients will be screened for HF risk factors using electronic medical records of participating family physicians to identify patients with potentially undiagnosed HF. Participants will then undergo a diagnostic evaluation using a blood sample for a hormone specific to the heart, the natriuretic peptide or NT-proBNP; if elevated, a portable cardiac ultrasound (ECHO) with artificial intelligence (AI) interpretation will be done; both NT-proBNP and ECHO are required for diagnosis in patients with signs and symptoms suggestive of HF. This screening ECHO coupled with AI reading from Us2.ai provides a fast, reliable, and inexpensive report, which is particularly important in our context, where waiting lists for such examinations can reach up to one year.

ELIGIBILITY:
Inclusion Criteria:

Male or female ≥40 years of age informed consent and at least two additional risk factors for HF: coronary artery disease [either a previous documented type 1 myocardial infarction or coronary artery bypass grafting or percutaneous coronary intervention or documented stenosis or an epicardial coronary artery (50% left main stem or >70% left anterior descending, circumflex or right coronary artery) diabetes type 1 or type 2, persistent or permanent atrial fibrillation, previous ischemic or embolic stroke peripheral arterial disease (previous surgical or percutaneous revascularization or documented stenosis >50% of major peripheral arterial vessel), chronic kidney disease (estimated glomerular filtration rate <60mL/min/1.73m2 or eGFR 60-90mL/min/1.73m2 and UACR >300mg/g), regular loop diuretic use for >30 days within 12 months COPD (evidenced by one of the following: PFTs showing airway obstruction diagnosis by respiratory physician CT scan reporting presence of emphysema, or treatment with national guideline COPD therapy).

Exclusion Criteria:

Inability to give informed consent e.g., due to significant cognitive impairment, previous diagnosis of heart failure (this is any diagnosis of heart failure with any ejection fraction of any cause) renal replacement therapy, anyone who, in the investigators' opinion, is not suitable to participate in the trial for other reasons e.g., a diagnosis which may compromise survival over the study period.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-11-20 (Actual); Primary Completion 2024-11-20 (Actual); Study Completion 2024-11-20 (Actual)

PRIMARY OUTCOMES:
Primary endpoint | 6 months
  In both arms the diagnosis of HF will be determined by the occurrence of one or more of the following (defined in Appendix 4):
  * An outpatient diagnosis of heart failure according to the ESC 2021 Heart Failure Guidelines.
  * Outpatient heart failure visit.
  * Urgent heart failure visit.
  * Heart failure hospitalisation.

SECONDARY OUTCOMES:
Secondary endpoints | 6 months
  Diagnosis of HFrEF within 6 months.
  • Patients diagnosed with HFrEF receiving GDMT within 6 months. Guideline-directed medical therapy is defined as simultaneously receiving the 4 drugs with a Class I guideline recommendation for HFrEF (unless not tolerated or contraindicated): Angiotensin receptor neprilysin inhibitor, beta blockers, mineralocorticoid receptor antagonists, sodium-glucose cotransporter-2 inhibitors.

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - University of British Columbia, Vancouver, British Columbia
  - Montreal Heart Institute, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No